CLINICAL TRIAL: NCT01425840
Title: Efficacy of Liposome Lidocaine Gel for Topical Anesthesia in the Palatal Mucosa
Brief Title: Liposomal Lidocaine Gel for Oral Topical Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 112/2007
Record Dates: First submitted 2011-08-24; First posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Anesthesia
Keywords: Lidocaine,; liposome encapsulation,; topical anesthesia,; palatal mucosa
MeSH Terms: interventions — Lidocaine; Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liposomal lidocaine, topical anesthesia (Experimental): Efficacy of Liposomal lidocaine in topical anesthesia.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — 100 mg of the following formulations: Liposome-encapsulated 2,5% and 5% lidocaine gel, liposome placebo gel and 2.5% lidocaine and 2.5% prilocaine cream were applied once during 5 minutes.
  Other Names: Topical anesthesia in the palatal mucosa

SUMMARY:
This blinded cross-over study aimed to evaluate the efficacy of topical liposome-encapsulated lidocaine on oral mucosa.

DETAILED DESCRIPTION:
This blinded cross-over study aimed to evaluate the efficacy of topical liposome-encapsulated 2,5 and 5% lidocaine gel formulations on the palatal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Volunteers were free from cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and haematological diseases, psychiatric disorders and allergy to local anesthetics

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The efficacy of topical anesthetics on the oral mucosa. | 10 seconds
  The topical formulations were kept in the palatal mucosa during 2 min. The efficacy of the topical formulations was assessed after a pinprick and a local anesthetic injection on the application site.

CONTACTS AND LOCATIONS:
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Result] Franz-Montan M, de Paula E, Groppo FC, Silva AL, Ranali J, Volpato MC. Liposomal delivery system for topical anaesthesia of the palatal mucosa. Br J Oral Maxillofac Surg. 2012 Jan;50(1):60-4. doi: 10.1016/j.bjoms.2010.10.018. Epub 2010 Nov 23. PMID 21106282